CLINICAL TRIAL: NCT02056405
Title: Effect of Mosapride on Postoperative Ileus in Patients Undergoing Colorectal Surgery
Acronym: ILEUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2104
Record Dates: First submitted 2014-01-31; First posted 2014-02-06 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Ileus
Keywords: Postoperative Ileus; Mosapride; Colorectal laparoscopic surgery; Prolonged postoperative ileus
MeSH Terms: interventions — mosapride; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo arm: intake of placebo (Lactose). 1 pill of the same characteristics as Mosapride every 8 hs with 30 ml tap water. This will begin on postoperative day 1 until discharge from Hospital or unacceptable toxicity develops.
  Interventions: Drug: Placebo
- Mosapride (Active Comparator): Mosapride arm: intake of active drug (Mosapride). 15 mg per day divided into 3 oral intakes of 5 mg each (1 pill of Mosapride every 8 hs with 30 ml tap water). This treatment will begin on postoperative day 1 until discharge from Hospital or unacceptable toxicity develops.
  Interventions: Drug: Mosapride

INTERVENTIONS:
Drug: Mosapride — 15 mg per day divided into 3 oral intakes of 5 mg each (1 pill of Mosapride every 8 hs with 30 ml tap water). This treatment will begin on postoperative day 1 until discharge from Hospital or unacceptable toxicity develops.
  Other Names: Mosar
  Arms: Mosapride
Drug: Placebo — 1 pill of the same characteristics as Mosapride every 8 hs with 30 ml tap water. This will begin on postoperative day 1 until discharge from Hospital or unacceptable toxicity develops.
  Other Names: Lactose
  Arms: Placebo

SUMMARY:
Postoperative Ileus is defined as the transient postoperative functional inhibition of propulsive bowel activity. The ethiology of this process can best be described as multifactorial. In its pathogenesis different mechanisms are involved such as hormones and neuropeptides, inflammation, narcotics and the Autonomic nervous system. Is one of the most common causes of prolonged hospital stays after abdominal surgery, thereby increasing health-care resource utilization. More importantly, it causes patient discomfort in the form of nausea, vomiting, and stomach cramps. It has a variable duration but is usually solved in 3 to 4 days. Prolonged Ileus is associated with postoperative complications like an increase on urinary and pulmonary infections, profound venous thrombosis and wound-site complications.

Mosapride is a prokinetic agent that acts as a selective serotonin agonist (5- HT4) that facilitates acetylcholine release from the intrinsic plexus. This accelerates gastric emptying and propulsive peristaltic movements on the lower intestines. Mosapride has no action over the central nervous system therefore the lesser side effects like cardiac arrhythmias and extrapyramidal symptoms. For being a safer drug we chose it to be the center of our research.

Two randomized controlled trials studied Mosapride concluding it shortens PI after colorectal surgery. However these trials took place on specific populations (Orientals) with less than 50 patients and only one of them included laparoscopic treatment specifically. Also the end point of these studies didn't consider the impact of PI over hospital stay or costs to the health system.

We therefore decided to conduct a prospective randomized study in patients undergoing laparoscopic colorectal surgery for colon cancer. The patients will be randomized to receive treatment or placebo after surgery. With this study we intend to prove that patients treated with mosapride immediately after surgery suffer from shorter postoperative ileus with earlier oral intake and shorter hospital stay.

The primary aim of the trial is to assess the effectiveness of the use of Mosapride in shortening the duration of the Postoperative ileus in patients undergoing colorectal laparoscopic surgery. The trial hypothesis is that the standardized use of Mosapride immediately after colorectal laparoscopic surgery is safe and accelerates the recovery of propulsive bowel activity, thereby shortening postoperative ileus and hospital stay.

DETAILED DESCRIPTION:
Methods. Design. Design A randomized controlled trial, triple blind with placebo. Study population Patients undergoing laparoscopic colorectal surgery. Italian Hospital of Buenos Aires. Argentina.

Inclusion and exclusion criteria

Participants will be eligible provided they are at least 18 years of age and under 85, are about to undergo colonic or upper rectum surgery with the diagnose of cancer o malignant polyp. People will be excluded if:

* They refuse to participate from the trial or the process of informed consent
* Have known allergies or hypersensitivity to Mosapride or lactose (used for placebo)
* Patients with ascites, hepatic metastases or carcinomatosis
* Patients who cannot receive Non-steroidal anti-inflammatory drugs
* Pregnancy or women at a fertile age who do not use double contraceptive agents
* Patients with conversion to laparotomy
* Patients with a Rectal tumor beneath 11 cm requiring low or ultralow rectal resection
* Patients with an stoma or who underwent simultaneous resection of other organs

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years old
* Underwent colonic or upper rectum laparoscopic surgery with diagnose of cancer or malignant polyp
* Were operated on Italian Hospital of Buenos Aires

Exclusion Criteria:

* They refuse to participate from the trial or the process of informed consent
* Have known allergies or hypersensitivity to Mosapride or lactose (used for placebo)
* Patients with ascites, hepatic metastases or carcinomatosis
* Patients who cannot receive Non-steroidal anti-inflammatory drugs
* Pregnancy or women at a fertile age who do not use double contraceptive agents
* Patients with conversion to laparotomy
* Patients with a Rectal tumor beneath 11 cm requiring low or ultralow rectal resection
* Patients with an derivative stoma or who underwent simultaneous resection of other organs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of days after Surgery until the recovery of bowel movement | 1 to 5 days after surgery
  Effect of the administration of mosapride on the immediate postoperative on the recovery of bowel movements.

SECONDARY OUTCOMES:
Number of patients to develop adverse reactions to Mosapride | 1 to 5 days after surgery
  To evaluate the safety of the administration of Mosapride after colorectal laparoscopic surgery.

OTHER OUTCOMES:
Number of days of Hospital stay after surgery. | 18 months (end of protocol)
  To assess the effect of Mosapride on the reduction of Hospital stay days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Vaccaro, MD, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Italian Hospital of Buenos Aires, Buenos Aires, State Capital, Argentina

REFERENCES:
- [Background] Toyomasu Y, Mochiki E, Morita H, Ogawa A, Yanai M, Ohno T, Fujii T, Tsutsumi S, Asao T, Kuwano H. Mosapride citrate improves postoperative ileus of patients with colectomy. J Gastrointest Surg. 2011 Aug;15(8):1361-7. doi: 10.1007/s11605-011-1567-x. Epub 2011 May 24. PMID 21607794
- [Background] Narita K, Tsunoda A, Takenaka K, Watanabe M, Nakao K, Kusano M. Effect of mosapride on recovery of intestinal motility after hand-assisted laparoscopic colectomy for carcinoma. Dis Colon Rectum. 2008 Nov;51(11):1692-5. doi: 10.1007/s10350-008-9407-0. Epub 2008 Jun 27. PMID 18584249
- [Background] Seta ML, Kale-Pradhan PB. Efficacy of metoclopramide in postoperative ileus after exploratory laparotomy. Pharmacotherapy. 2001 Oct;21(10):1181-6. doi: 10.1592/phco.21.15.1181.33888. PMID 11601663
- [Background] Davidson ED, Hersh T, Brinner RA, Barnett SM, Boyle LP. The effects of metoclopramide on postoperative ileus. A randomized double-blind study. Ann Surg. 1979 Jul;190(1):27-30. doi: 10.1097/00000658-197907000-00006. PMID 582360
- [Background] Furness JB, Costa M. Adynamic ileus, its pathogenesis and treatment. Med Biol. 1974 Apr;52(2):82-9. No abstract available. PMID 4365867
- [Background] Jepsen S, Klaerke A, Nielsen PH, Simonsen O. Negative effect of Metoclopramide in postoperative adynamic ileus. A prospective, randomized, double blind study. Br J Surg. 1986 Apr;73(4):290-1. doi: 10.1002/bjs.1800730414. PMID 3516299
- [Background] Tollesson PO, Cassuto J, Rimback G, Faxen A, Bergman L, Mattsson E. Treatment of postoperative paralytic ileus with cisapride. Scand J Gastroenterol. 1991 May;26(5):477-82. doi: 10.3109/00365529108998569. PMID 1871540
- [Background] Brown TA, McDonald J, Williard W. A prospective, randomized, double-blinded, placebo-controlled trial of cisapride after colorectal surgery. Am J Surg. 1999 May;177(5):399-401. doi: 10.1016/s0002-9610(99)00071-9. PMID 10365879